CLINICAL TRIAL: NCT07190027
Title: Prospective Randomized Controlled Trial of Immunodynamics-Guided Optimization of Individualized Immunochemotherapy Infusion Timing in Driver Gene-Negative Advanced Non-Small Cell Lung Cancer
Brief Title: Immunodynamics-Guided Optimization of Individualized Immunochemotherapy in Advanced Driver-Negative NSCLC: A Randomized Trial
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: First Affiliated Hospital of Wenzhou Medical University (Other)
Responsible Party: Principal Investigator, Liang bin, Clinical Investigator, First Affiliated Hospital of Wenzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY2025-309
Record Dates: First submitted 2025-09-10; First posted 2025-09-24 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Advanced Non-Small Cell Lung Cancer (NSCLC)
Keywords: Non-Small Cell Lung Cancer (NSCLC); Driver Gene-Negative NSCLC; Immunochemotherapy Sequencing; Individualized Infusion Timing; Immune Dynamics
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Drug Therapy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Arm 2: Fixed Delay Group (Experimental): Patients receive standard chemotherapy on Day 1 of each 21-day cycle. The PD-1 inhibitor is administered with a fixed delay, on Day 4 (3 days after chemotherapy). Combination treatment is given for 4 cycles, followed by PD-1 inhibitor maintenance until disease progression, unacceptable toxicity
  Interventions: Drug: Arm 2：Fixed Delay Group
- Arm 1: Standard Synchronous Group (Experimental): Patients receive standard chemotherapy and PD-1 inhibitor concurrently on Day 1 of each 21-day cycle. After 4 cycles of combination therapy, patients continue PD-1 inhibitor maintenance until progression
  Interventions: Drug: Arm 1： Standard Synchronous Group
- Arm 3: Individualized Delay Group (Experimental): Patients receive chemotherapy on Day 1 of each 21-day cycle. From Day 2 to Day 5, peripheral blood immunodynamic markers (e.g., CD8⁺PD-1⁺ T cells, MDSCs, Tregs, cytokines) are monitored daily. The PD-1 inhibitor is administered at the optimal time when predefined immunodynamic criteria are met, or on Day 6 if criteria are not met. After 4 cycles of combination therapy, patients continue PD-1 inhibitor maintenance until progression
  Interventions: Drug: Arm 3： Individualized Delay Group

INTERVENTIONS:
Drug: Arm 1： Standard Synchronous Group — Arm 1: Concurrent PD-1 + Chemotherapy (Standard Synchronous Group) Participants in this group will receive PD-1 inhibitor and chemotherapy on the same day (D1) during each treatment cycle.
  Other Names: Concurrent PD-1 + Chemotherapy
  Arms: Arm 1: Standard Synchronous Group
Drug: Arm 2：Fixed Delay Group — Fixed Delay Arm Delayed PD-1 + Chemo PD-1 inhibitor (e.g., Sintilimab/Keytruda/Tislelizumab/Camrelizumab/Toripalimab/Nivolumab/Atezolizumab/Sugemalimab) Immune checkpoint inhibitor + Chemo (Day 3)
  Other Names: PD-1 Delayed Administration on D3 (Fixed Delay Group) Participants in this group will receive chemotherapy on D1 and then receive the PD-1 inhibitor on D3 of each cycle.
  Arms: Arm 2: Fixed Delay Group
Drug: Arm 3： Individualized Delay Group — Arm 3: Individualized PD-1 Timing Based on Immune Window Score (IWS) (Individualized Group) Participants in this group will receive chemotherapy on D1 and undergo daily immune monitoring (CD8⁺PD-1⁺ T cells, Treg, IFN-γ, NLR, ALC, CRP).
  Based on the immune window score (IWS):
  If IWS ≥ 2, PD-1 inhibitor will be administered the same day. If IWS = 1-1.5, dosing may be delayed to D3-D5 depending on immune recovery. If IWS remains 0 by D5, PD-1 inhibitor will be administered on D6 as fallback.
  Arms: Arm 3: Individualized Delay Group

SUMMARY:
The goal of this clinical trial is to evaluate whether individualized sequencing of immunotherapy and chemotherapy based on immune dynamics can improve treatment outcomes in adults with advanced non-small cell lung cancer (NSCLC) without driver gene mutations. This study will also assess the safety and feasibility of different infusion strategies.

The main questions it aims to answer are:

Does optimizing the timing of PD-1 inhibitor infusion relative to chemotherapy improve the objective response rate (ORR)?

Does individualized infusion sequencing enhance progression-free survival (PFS) compared to standard or fixed-delay administration?

What safety concerns or immune-related adverse events occur with different infusion timing strategies?

Researchers will compare three treatment strategies:

Group A (Standard Concurrent Group): Immunotherapy and chemotherapy administered on the same day (D1).

Group B (Fixed Delay Group): Chemotherapy on D1, followed by PD-1 inhibitor infusion on Day 3.

Group C (Individualized Delay Group): Chemotherapy on D1, and PD-1 inhibitor infusion scheduled on D2-D6 based on daily immune monitoring.

Participants will:

Receive a PD-1 inhibitor (e.g., sintilimab, pembrolizumab, camrelizumab) combined with platinum-based chemotherapy.

Attend clinic visits for regular immune monitoring, imaging assessments, and safety checks during each treatment cycle.

Undergo blood tests to evaluate immune biomarkers (e.g., CD8⁺PD-1⁺ T cells, MDSC, Treg、IFN-γ、NLR、ALC、CRP) to guide individualized treatment decisions.

DETAILED DESCRIPTION:
Detailed Description

This study is a prospective, randomized, open-label, multicenter exploratory clinical trial designed to evaluate the efficacy and safety of immunodynamics-guided optimization of chemoimmunotherapy scheduling in patients with advanced non-small cell lung cancer (NSCLC) without targetable driver mutations. The trial specifically investigates whether individualized scheduling of PD-1 inhibitor infusion, guided by dynamic immune monitoring, can improve antitumor activity compared with standard synchronous or fixed-delay administration.

Rationale and Background

For patients with metastatic NSCLC lacking EGFR, ALK, or other approved targetable alterations, chemoimmunotherapy has become the standard first-line treatment. However, clinical outcomes remain heterogeneous, and not all patients benefit equally. Preclinical and translational evidence suggests that the timing of immune checkpoint blockade relative to chemotherapy exposure may significantly influence immune response, tumor microenvironment remodeling, and overall treatment efficacy. Immunodynamics-the dynamic assessment of immune status during therapy-offers a novel approach to guide individualized administration of immunotherapy, potentially enhancing efficacy while maintaining safety.

Study Objectives

Primary Objective: To compare the objective response rate (ORR) among three treatment arms:

Arm A: Standard synchronous administration of chemotherapy and PD-1 inhibitor.

Arm B: Fixed-delay administration, with PD-1 inhibitor given three days after chemotherapy.

Arm C: Individualized-delay administration, where PD-1 inhibitor infusion timing (Day 2-6) is determined by peripheral blood immunodynamic markers.

Secondary Objectives: To evaluate progression-free survival (PFS), overall survival (OS), disease control rate (DCR), duration of response (DOR), safety, and incidence of immune-related adverse events (irAEs).

Exploratory Objectives: To explore the relationship between immune scheduling and peripheral immune dynamics (CD8⁺PD-1⁺ T cells, myeloid-derived suppressor cells [MDSCs], Tregs, cytokines, etc.), as well as the predictive value of these markers for therapeutic outcomes.

Study Design

A total of 246 eligible patients with untreated metastatic, driver gene-negative NSCLC will be randomized in a 1:1:1 ratio into Arms A, B, and C (82 patients per arm). Treatment will consist of four cycles of chemoimmunotherapy followed by PD-1 inhibitor maintenance until disease progression, unacceptable toxicity, or a maximum of 2 years.

Arm A (Standard Synchronous): Chemotherapy and PD-1 inhibitor administered on Day 1 of each cycle.

Arm B (Fixed-Delay): Chemotherapy on Day 1; PD-1 inhibitor on Day 4.

Arm C (Individualized-Delay): Chemotherapy on Day 1; immune markers (CD8⁺PD-1⁺ T cells, MDSCs, Tregs, ± cytokines) measured on Days 2-5; PD-1 inhibitor administered when immunodynamic criteria are met, or on Day 6 as default.

Treatment cycles will repeat every 3 weeks. Imaging will be performed every 6 weeks during the first 48 weeks, then every 9 weeks, using RECIST v1.1 criteria. Patients will be followed for safety and survival after treatment discontinuation.

Endpoints

Primary Endpoint: Objective response rate (ORR) assessed by independent radiologic review committee (IRC).

Secondary Endpoints: PFS, OS, DCR, DOR, safety, incidence and severity of irAEs and treatment-related adverse events.

Exploratory Endpoints: Dynamic immune monitoring parameters, association between immune recovery patterns and clinical outcomes, correlation of PD-L1 expression and immune biomarkers, and exploratory ctDNA analyses if feasible.

Statistical Considerations

The study is powered to detect clinically meaningful improvements in ORR. Stratified CMH tests will be used for ORR comparisons. Kaplan-Meier methods and Cox proportional hazards models will be applied for time-to-event endpoints (PFS, OS, DOR). Exploratory analyses will examine associations between immunodynamic markers and outcomes, and predictive biomarker models will be developed. Safety analyses will summarize adverse events by frequency, grade, and relatedness.

Significance

This trial represents the first randomized study to prospectively test immunodynamics-guided optimization of immunochemotherapy scheduling in NSCLC. By integrating real-time immune monitoring into treatment decision-making, the study aims to generate evidence for precision timing of PD-1 inhibitor administration, potentially enhancing treatment efficacy and safety. Results from this study may inform future clinical practice and contribute to individualized immunotherapy strategies in lung cancer and beyond.

ELIGIBILITY:
Inclusion Criteria:

Participants must meet all of the following criteria:

Voluntarily agree to participate, sign the informed consent form (ICF), and be able to comply with the study procedures.

Age ≥18 years and ≤75 years at enrollment, both male and female participants are eligible.

Histologically or cytologically confirmed stage IV non-small cell lung cancer (NSCLC) based on the AJCC 8th edition; if mixed histology exists, classification must be based on the predominant histologic component. Presence of small-cell histology excludes eligibility.

Negative for actionable driver mutations: no EGFR mutations, ALK rearrangements, or ROS1 fusions. For other targetable alterations (e.g., BRAF V600E, NTRK1/2/3 fusions, MET exon 14 skipping, RET rearrangements), patients are excluded if FDA- or NMPA-approved targeted therapies are available.

Note: Genetic testing can be conducted locally or via a central laboratory. Pre-existing valid reports are acceptable.

Estimated life expectancy ≥3 months. At least one measurable lesion per RECIST v1.1 confirmed by IRC; irradiated lesions are not considered measurable unless unequivocal progression is demonstrated.

ECOG performance status of 0 or 1. No prior systemic therapy for advanced/metastatic NSCLC, except adjuvant or neoadjuvant chemotherapy if the last dose was ≥6 months before recurrence.

Adequate organ and bone marrow function within 14 days prior to randomization:

ANC ≥ 1.5 × 10⁹/L Platelets ≥ 100 × 10⁹/L Hemoglobin ≥ 90 g/L Serum creatinine ≤ 1.5 × ULN or creatinine clearance ≥ 50 mL/min (Cockcroft-Gault formula) Total bilirubin ≤ 1.5 × ULN (≤3 × ULN for Gilbert's syndrome) AST/ALT ≤ 2.5 × ULN (≤5 × ULN if liver metastases) INR and APTT ≤ 1.5 × ULN unless on therapeutic anticoagulation LVEF ≥ 50% by echocardiography or MUGA Female patients of childbearing potential must test negative for pregnancy within 14 days before enrollment and agree to use effective contraception from ICF signing until 180 days after the last dose. Male participants must also agree to effective contraception during the same period.

Exclusion Criteria:

Participants meeting any of the following are excluded:

Prior thoracic radiotherapy >30 Gy within 6 months before first dose. Palliative radiotherapy within 7 days before first dose. Requirement for concurrent anti-tumor therapy during the study. Uncontrolled or symptomatic pleural, pericardial, or peritoneal effusions requiring repeated drainage.

Brainstem, leptomeningeal, spinal cord metastases, or cord compression.

Active CNS metastases or carcinomatous meningitis. Treated, stable brain metastases are allowed if:

Clinically stable ≥2 weeks, No evidence of progression, Off corticosteroids ≥3 days prior to treatment initiation. Previous treatment with immune checkpoint inhibitors (PD-1/PD-L1, CTLA-4, etc.), immune agonists, or cellular immunotherapies.

Use of traditional Chinese medicines or immunomodulatory drugs with anti-cancer activity within 2 weeks before first dose.

Systemic corticosteroids (>10 mg prednisone equivalent/day) or other immunosuppressants within 2 weeks prior to first dose.

Uncontrolled systemic infection, unexplained fever >38.5°C, or IV antibiotic use >7 days within 2 weeks prior to first dose.

History of other malignancies within the past 5 years, except adequately treated cervical carcinoma in situ, basal/squamous cell skin cancer, localized thyroid papillary carcinoma, prostate cancer in remission, or DCIS after curative surgery.

Active or history of autoimmune disease, including but not limited to: autoimmune hepatitis, interstitial lung disease, uveitis, colitis, hepatitis, pituitary inflammation, vasculitis, nephritis, hyperthyroidism, or hypothyroidism.

Controlled hypothyroidism with hormone replacement is eligible. Vitiligo, alopecia, type 1 diabetes, resolved childhood asthma, or mild psoriasis without systemic therapy are allowed.

Clinically significant pulmonary diseases: e.g., steroid-requiring pneumonitis, drug-induced pneumonitis, or moderate-to-severe COPD.

Major surgery within 4 weeks prior to first dose or unresolved surgical wounds.

Significant cardiovascular diseases, including:

MI, unstable angina, stroke, or TIA within 6 months Arterial thromboembolism within 6 months DVT, PE, or severe thrombosis within 3 months Uncontrolled hypertension (SBP ≥160 mmHg or DBP ≥100 mmHg) Myocarditis or NYHA III-IV heart failure History of allogeneic HSCT or organ transplantation (except corneal).

≥ Grade 2 peripheral neuropathy per CTCAE v5.0. Active tuberculosis or suspected TB not ruled out. Positive HIV antibody; active syphilis or untreated positive non-treponemal antibody; uncontrolled HBV/HCV infection per protocol definition.

Live vaccine administration within 30 days before first dose or planned during study.

History of severe hypersensitivity to monoclonal antibodies, PD-1 agents, pemetrexed, carboplatin, or premedications.

Concurrent participation in another interventional clinical trial or use of other investigational products/devices within 4 weeks prior to first dose.

History of drug/alcohol abuse or uncontrolled psychiatric disorders interfering with compliance.

Any other condition judged by the investigator as inappropriate for study participation.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 246 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From baseline until disease progression, death, or completion of treatment, whichever occurs first, up to approximately 36 months.
  The proportion of participants who achieve a complete response (CR) or partial response (PR) based on RECIST v1.1 criteria, as assessed by investigators. Imaging assessments will be performed every 6-8 weeks during treatment, and responses will be confirmed at least 4 weeks after initial documentation.

SECONDARY OUTCOMES:
PFS | From baseline until documented disease progression or death, up to approximately 36 months.
  PFS is defined as the time from the start of treatment until disease progression as assessed by RECIST v1.1 criteria or death from any cause, whichever occurs first. Imaging assessments will be performed every 6-8 weeks.
Overall Survival (OS) | From baseline until death from any cause, up to approximately 48 months.
  OS is defined as the time from the start of treatment until death from any cause. Participants alive at the time of analysis will be censored at the last date known to be alive.
Incidence of Immune-Related Adverse Events (irAEs) | From baseline through 90 days after the last dose of study treatment, up to approximately 36 months.
  The percentage of participants experiencing any grade immune-related adverse events, as defined by CTCAE v5.0, including but not limited to dermatitis, colitis, pneumonitis, hepatitis, and endocrinopathies.
Incidence of Treatment-Related Adverse Events (TRAEs) | From baseline through 90 days after the last dose of study treatment, up to approximately 36 months.
  The percentage of participants experiencing any grade treatment-related adverse events, assessed by investigators and graded according to CTCAE v5.0.

OTHER OUTCOMES:
Proportion and Activation Status of CD8⁺PD-1⁺ T Cells | From baseline to the end of treatment, up to 36 months.
  Flow cytometry will be used to measure the proportion and activation status of CD8⁺ T cells expressing PD-1 in peripheral blood. The dynamic changes in CD8⁺PD-1⁺ T cells will be analyzed in relation to treatment response and immune modulation.
Proportion of Regulatory T Cells (Treg) | From baseline to the end of treatment, up to 36 months.
  Flow cytometry will be used to assess the percentage and absolute count of CD4⁺CD25⁺FoxP3⁺ regulatory T cells (Treg) in peripheral blood, and their association with treatment efficacy and immune-related adverse events.
Proportion of Myeloid-Derived Suppressor Cells (MDSC) | From baseline to the end of treatment, up to 36 months.
  Flow cytometry will measure the proportion of MDSCs, including polymorphonuclear-MDSCs (PMN-MDSC) and monocytic-MDSCs (M-MDSC), in peripheral blood. The relationship between MDSC levels and therapeutic response will be analyzed.
Neutrophil-to-Lymphocyte Ratio (NLR) | From baseline to the end of treatment, up to 36 months.
  NLR will be calculated from routine complete blood counts. The correlation between NLR dynamics and treatment response, progression-free survival (PFS), and immune-related adverse events will be assessed.
Absolute Lymphocyte Count (ALC) | From baseline to the end of treatment, up to 36 months.
  ALC will be obtained from complete blood counts and analyzed as an exploratory biomarker for immune activation and treatment outcomes.
Serum Interferon Gamma (IFN-γ) Concentration | From baseline to the end of treatment, up to 36 months.
  Serum IFN-γ levels will be quantified by ELISA to assess immune activation status and their predictive value for treatment response.
Serum C-Reactive Protein (CRP) Level | From baseline to the end of treatment, up to 36 months.
  CRP levels will be measured using immunoturbidimetry or high-sensitivity assays to evaluate systemic inflammatory status and its association with treatment efficacy and immune-related adverse events.

IPD SHARING:
Plan to Share IPD: No